CLINICAL TRIAL: NCT03240939
Title: A Randomized, Open Label, Single Dose, Two-way Crossover Clinical Trial to Investigate the Pharmacokinetics and Safety/Tolerability of YY-201 in Comparison to Dutasteride and Tadalafil Administered in Healthy Male Volunteer
Brief Title: Pharmacokinetics and Safety/Tolerability of YY-201 in Comparison to Dutasteride and Tadalafil
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuyu Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: YY-201_PK
Record Dates: First submitted 2017-04-24; First posted 2017-08-07 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-05

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Dutasteride; Tadalafil
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Dutasteride; Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dutasteride&Tadalafil (Active Comparator): Dutasteride 0.5 mg capsule and Tadalafil 5 mg Tablet, single dose
  Interventions: Drug: Dutasteride 0.5 mg; Drug: Tadalafil 5 mg
- YY-201 (Experimental): YY-201 capsule, singe dose
  Interventions: Drug: YY-201

INTERVENTIONS:
Drug: Dutasteride 0.5 mg — single dose
  Arms: Dutasteride&Tadalafil
Drug: Tadalafil 5 mg — single dose
  Arms: Dutasteride&Tadalafil
Drug: YY-201 — single dose
  Arms: YY-201

SUMMARY:
A randomized, open label, single dose, two-way crossover clinical trial to investigate the pharmacokinetics and safety/tolerability of YY-201 in comparison to Dutasteride and Tadalafil administered in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Age 19 to 45 years
* BMI score 19 kg/m2 to 28 kg/m2
* SBP < 140 mmHg and ≤ 90 mmHg or DBP < 90 mmHg and ≥ 50 mmHg
* Eligible according to the laboratory results of hematology, blood chemistry and urinalysis
* Voluntarily signed the informed consent form

Exclusion Criteria:

* Gastrointestinal diseases or surgery which may affect absorption of the investigational products within 6 months
* History of hypersensitivity
* history of Cardiovascular disease
* History of degenerative Retina disease
* Lactose intolerance
* Medical history of vision loss
* Clinically significant disorders of allergy, drug hypersensitivity reaction, hepatobiliary system, kidney, neurology, respiratory, hemato-oncology, endocrine, dermatology, urology, ophthalmology, psychiatry, musculo-skeletal system, immunology, otorhinolaryngology, and cardiovascular system
* Donated whole blood (transfusion, apheresis etc..) within 60 days
* Participated and administered the investigational products in other clinical trial within 90 days
* Taking drugs which may affect Clinical trial within 30 days
* Smoked more than 10 cigarettes a day for past 30 days
* Excessive alcohol consumption (> 3 units/week, 1 unit)
* Taking food which may affect Clinical trial within 7 days
* Positive result from Urinary test
* Positive result from Serum test
* Clinically significant disorders result from Electrocardiography test
* Not eligible due to investigator's judgments

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2017-07-07 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
Cmax | Day 1 0 hour (pre-dose), 0.5 hour, 1hour, 1.5hour, 2hour, 2.5hour, 3hour, 3.5hour, 4hour, 5hour, 6hour, 8hour, 12hour, 24hour(Day 2), 32 hour, 48hour(Day 3), 72hour(Day 4), 96hour(Day 5), 144hour(Day 7), 192hour(Day 9), 240hour(Day 11)
  "Peak Plasma Concentration" of Dutasteride, tadalafil

SECONDARY OUTCOMES:
Tmax | Day 1 0 hour (pre-dose), 0.5 hour, 1hour, 1.5hour, 2hour, 2.5hour, 3hour, 3.5hour, 4hour, 5hour, 6hour, 8hour, 12hour, 24hour(Day 2), 32 hour, 48hour(Day 3), 72hour(Day 4), 96hour(Day 5), 144hour(Day 7), 192hour(Day 9), 240hour(Day 11)
  Time at which the maximum concentration of Dutasteride, Tadalafil
t1/2β | Day 1 0 hour (pre-dose), 0.5 hour, 1hour, 1.5hour, 2hour, 2.5hour, 3hour, 3.5hour, 4hour, 5hour, 6hour, 8hour, 12hour, 24hour(Day 2), 32 hour, 48hour(Day 3), 72hour(Day 4), 96hour(Day 5), 144hour(Day 7), 192hour(Day 9), 240hour(Day 11)
  half-life
AUCinf | Day 1 0 hour (pre-dose), 0.5 hour, 1hour, 1.5hour, 2hour, 2.5hour, 3hour, 3.5hour, 4hour, 5hour, 6hour, 8hour, 12hour, 24hour(Day 2), 32 hour, 48hour(Day 3), 72hour(Day 4), 96hour(Day 5), 144hour(Day 7), 192hour(Day 9), 240hour(Day 11)
  area under the plasma concentration versus time curve of Dutasteride, Tadalafil

CONTACTS AND LOCATIONS:
Overall Officials: Hyeong-Seok Lim, M.D.,Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea